CLINICAL TRIAL: NCT02915302
Title: Safety and Immunogenicity of Fluzone® Quadrivalent Vaccine Administered to Healthy Children 6 to < 36 Months of Age
Brief Title: Safety and Immunogenicity of Fluzone® Quadrivalent Vaccine Administered to Healthy Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRC88; U1111-1143-9273 (Other: WHO)
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus vaccine; Fluzone® Quadrivalent Influenza Vaccine (No Preservative)
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone Quadrivalent Vaccine, 0.25-mL (Active Comparator): Participants received a 0.25-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. For participants for whom 2 doses of influenza vaccine were recommended per ACIP guidance, a second 0.25-mL dose of Fluzone Quadrivalent vaccine was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, No Preservative
- Fluzone Quadrivalent Vaccine, 0.5-mL (Experimental): Participants received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. For participants for whom 2 doses of influenza vaccine were recommended per ACIP guidance, a second 0.5-mL dose of Fluzone Quadrivalent vaccine was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, No Preservative

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine, No Preservative — 0.25-mL (Pediatric Dose), Intramuscular (2016-2017 formulation)
  Other Names: Fluzone® Quadrivalent Influenza Vaccine
  Arms: Fluzone Quadrivalent Vaccine, 0.25-mL
Biological: Fluzone Quadrivalent vaccine, No Preservative — 0.5-mL, Intramuscular (2016-2017 formulation)
  Other Names: Fluzone® Quadrivalent Influenza Vaccine
  Arms: Fluzone Quadrivalent Vaccine, 0.5-mL

SUMMARY:
The aim of the study was to describe the safety and immunogenicity of a 0.5-mL dose (15 μg hemagglutinin [HA] per strain) of Fluzone Quadrivalent vaccine in children 6 to <36 months of age.

Primary objective:

* To compare the rate of any fever (temperature ≥100.4 degrees Fahrenheit [38.0 degrees Celsius) following a 0.5-mL dose of Fluzone Quadrivalent vaccine to that following a 0.25-mL dose of Fluzone Quadrivalent vaccine during the 7 days after either vaccination (Dose 1 and Dose 2 combined) in participants 6 to < 36 months of age.

Secondary objective:

* To compare antibody responses induced by a 0.5-mL dose of Fluzone Quadrivalent vaccine to those induced by a 0.25-mL dose of Fluzone Quadrivalent vaccine as assessed by geometric mean titer (GMT) ratios and seroconversion rate differences after the final vaccination in participants 6 to < 36 months of age.

Other objectives:

* To describe the safety of 2 different dose levels of the 2016-2017 formulation of Fluzone Quadrivalent vaccine in participants 6 to < 36 months of age.
* To describe the immunogenicity of 2 different dose levels of the 2016-2017 formulation of Fluzone Quadrivalent vaccine in participants 6 months to < 36 months of age.
* To submit available sera from approximately 30 participants to the Center for Biologics Evaluation and Research for further analysis by the World Health Organization, the Centers for Disease Control and Prevention, and the FDA to support formulation recommendations for subsequent influenza vaccines.

DETAILED DESCRIPTION:
All participants received 1 intramuscular dose of Fluzone Quadrivalent vaccine during Visit 1. For participants, for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP) guidance, a second dose of Fluzone Quadrivalent vaccine (of the same volume as the first dose) was administered during Visit 2 (28 days after Visit 1).

Solicited adverse event (AE) information was collected for 7 days after each vaccination, unsolicited AE information was collected from Visit 1 to Visit 2 or to Visit 3 for participants receiving 2 doses of study vaccine. Serious adverse event (SAE) information was collected for 28 days after each vaccination.

Immunogenicity was evaluated in a planned subset of 1600 randomly selected participants prior to vaccination on Day 0 (Visit 1) and at Day 28 after the final vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to < 36 months of age on the day of first study vaccination (study product administration).
* Born at full term of pregnancy (≥37 weeks) and/or with a birth weight ≥2.5 kg. Note: This inclusion criterion only applies to participants 6 to <12 months of age on the day of the first study visit.
* Informed consent form has been signed and dated by the parent(s) or guardian(s).
* Participant and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 30 days preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 30 days preceding the first trial vaccination, or planned receipt of any vaccine before Visit 2 for participants receiving 1 dose of influenza vaccine or Visit 3 for participants receiving 2 doses of influenza vaccine.
* Previous vaccination against influenza (in the 2016-2017 season) with either the trial vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of planned vaccination or febrile illness (temperature ≥100.4 degrees Fahrenheit [38.0 degrees Celsius]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as a natural or adopted child of either the Investigator or an employee with direct involvement in the proposed study.
* History of serious adverse reactions to any influenza vaccine.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1950 (Actual)
Dates: Start 2016-09-23; Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (32):
- United States (31):
  - Birmingham, Alabama
  - Harrisburg, Arkansas
  - Downey, California
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - Thornton, Colorado
  - Miami, Florida
  - Miami Beach, Florida
  - Meridian, Idaho
  - Bardstown, Kentucky
  - Metairie, Louisiana
  - Lincoln, Nebraska
  - Norfolk, Nebraska
  - Omaha, Nebraska
  - Syracuse, New York
  - Dayton, Ohio
  - Grove City, Ohio
  - Gresham, Oregon
  - Erie, Pennsylvania
  - Charleston, South Carolina
  - Tullahoma, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Layton, Utah
  - Orem, Utah
  - Provo, Utah
  - Roy, Utah
  - South Jordan, Utah
  - West Jordan, Utah
  - Burke, Virginia
- Anaheim, California, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Robertson CA, Mercer M, Selmani A, Klein NP, Jeanfreau R, Greenberg DP. Safety and Immunogenicity of a Full-dose, Split-virion, Inactivated, Quadrivalent Influenza Vaccine in Healthy Children 6-35 Months of Age: A Randomized Controlled Clinical Trial. Pediatr Infect Dis J. 2019 Mar;38(3):323-328. doi: 10.1097/INF.0000000000002227. PMID 30395011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 38 centers in the United States from 23 September 2016 to 02 January 2017.
Pre-assignment Details: A total of 1950 participants were randomized in the study.
Groups:
- Fluzone Quadrivalent Vaccine, 0.25-mL: Participants received a 0.25-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. For participants for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP) guidance, a second 0.25-mL dose of Fluzone Quadrivalent vaccine was administered at Day 28.
Period: Overall Study
Arm/Group | Fluzone Quadrivalent Vaccine, 0.25-mL | Fluzone Quadrivalent Vaccine, 0.5-mL
Started | 955 | 995
Vaccinated (Safety Analysis Set) | 949 | 992
Completed | 890 | 917
Not Completed | 65 | 78
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 20 | 27
Not completed — Lost to Follow-up | 19 | 22
Not completed — Withdrawal by Subject | 22 | 29
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed using the safety analysis set which included those participants who received at least 1 dose of study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone Quadrivalent Vaccine, 0.25-mL | Fluzone Quadrivalent Vaccine, 0.5-mL | Total
Number analyzed (Participants) | 949 | 992 | 1941
Age, Continuous [Mean (Standard Deviation); unit: Months] | 20.4 (8.75) | 20.5 (8.55) | 20.5 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 469 | 495 | 964
  Male | 480 | 497 | 977
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 206 | 221 | 427
  Not Hispanic or Latino | 731 | 763 | 1494
  Unknown or Not Reported | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 10 | 19
  Asian | 1 | 8 | 9
  Native Hawaiian or Other Pacific Islander | 4 | 5 | 9
  Black or African American | 178 | 195 | 373
  White | 717 | 725 | 1442
  More than one race | 36 | 43 | 79
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 949 | 992 | 1941

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Fever (Fever Rate) Following Vaccination With Fluzone Quadrivalent Vaccine
Description: Fever rate was defined as percentage of participants with fever (temperature >=100.4 degrees Fahrenheit [38.0 degrees Celsius]) following vaccination with Fluzone Quadrivalent vaccine.
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed using the safety analysis set. Here, 'Number of participants analyzed' = those participants with available data for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone Quadrivalent Vaccine, 0.25-mL | Fluzone Quadrivalent Vaccine, 0.5-mL
Number analyzed (Participants) | 893 | 930
percentage of participants | 11.31 [9.31 to 13.57] | 12.15 [10.12 to 14.42]
Statistical Analysis 1: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; Difference in fever rate was defined as the fever rate following a 0.5-mL dose of Fluzone Quadrivalent vaccine minus the fever rate following a 0.25-mL dose of Fluzone Quadrivalent vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper limit of the 2-sided 95% confidence interval (CI) of the difference in fever rate was <5%; Difference in Fever Rate = 0.84, 95% CI 2-sided [-2.13 to 3.80] — Fever rate: Fluzone Quadrivalent vaccine (0.5-mL vs. 0.25-mL)

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, B Yamagata lineage.
Time Frame: 28 days post-final vaccination
Population: Analysis was performed using Per-protocol (PP) analysis set which included participants who received at least 1 dose of study vaccine and had a valid post-vaccination serologic result for at least 1 strain without any protocol deviations. Here, 'Number Analyzed' = those participants with available data for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions [dil])
Arm/Group | Fluzone Quadrivalent Vaccine, 0.25-mL | Fluzone Quadrivalent Vaccine, 0.5-mL
Number analyzed (Participants) | 525 | 543
Titers (1/dilutions [dil])
  A/H1N1: number analyzed (Participants) | 520 | 539
  A/H1N1 | 214 [185 to 247] | 310 [271 to 354]
  A/H3N2: number analyzed (Participants) | 525 | 542
  A/H3N2 | 221 [191 to 256] | 332 [290 to 380]
  B Victoria: number analyzed (Participants) | 520 | 539
  B Victoria | 261 [227 to 299] | 348 [304 to 398]
  B Yamagata: number analyzed (Participants) | 524 | 543
  B Yamagata | 243 [213 to 277] | 349 [307 to 397]
Statistical Analysis 1: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For A/H1N1 strain, GMT ratio was defined as the GMT after 0.5 mL dose(s) of Fluzone Quadrivalent vaccine divided by the GMT after 0.25 mL dose(s) of Fluzone Quadrivalent vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the ratio of GMTs was >0.667; GMTs Ratio (A/H1N1) = 1.45, 95% CI 2-sided [1.19 to 1.77] — A/H1N1 strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)
Statistical Analysis 2: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For A/H3N2 strain, GMT ratio was defined as the GMT after 0.5 mL dose(s) of Fluzone Quadrivalent vaccine divided by the GMT after 0.25 mL dose(s) of Fluzone Quadrivalent vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the ratio of GMTs was >0.667; GMTs Ratio (A/H3N2) = 1.50, 95% CI 2-sided [1.23 to 1.83] — A/H3N2 strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)
Statistical Analysis 3: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For B Victoria lineage strain, GMT ratio was defined as the GMT after 0.5 mL dose(s) of Fluzone Quadrivalent vaccine divided by the GMT after 0.25 mL dose(s) of Fluzone Quadrivalent vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the ratio of GMTs was >0.667; GMTs Ratio (B Victoria lineage) = 1.33, 95% CI 2-sided [1.10 to 1.62] — B Victoria lineage strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)
Statistical Analysis 4: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For B Yamagata lineage strain, GMT ratio was defined as the GMT after 0.5 mL dose(s) of Fluzone Quadrivalent vaccine divided by the GMT after 0.25 mL dose(s) of Fluzone Quadrivalent vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the ratio of GMTs was >0.667; GMTs Ratio (B Yamagata lineage) = 1.44, 95% CI 2-sided [1.20 to 1.73] — B Yamagata lineage strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)

3. Secondary Outcome: Percentage of Participants With Seroconversion (Seroconversion Rate [SCR]) to Influenza Vaccine Antigens
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, B Yamagata lineage. SCR was defined as percentage of participants with either a pre-vaccination titer <10 (1/dil) and a post-final vaccination titer >=40 (1/dil), or a pre-vaccination titer >=10 (1/dil) and at least a four-fold increase in post-final vaccination titer.
Time Frame: 28 days post-final vaccination
Population: Analysis was performed using the PP analysis set. Here, 'Number Analyzed' = those participants with available data for specified categories.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone Quadrivalent Vaccine, 0.25-mL | Fluzone Quadrivalent Vaccine, 0.5-mL
Number analyzed (Participants) | 525 | 543
percentage of participants
  A/H1N1: number analyzed (Participants) | 470 | 483
  A/H1N1 | 78.9 [75.0 to 82.5] | 84.1 [80.5 to 87.2]
  A/H3N2: number analyzed (Participants) | 475 | 487
  A/H3N2 | 81.9 [78.1 to 85.3] | 86.2 [82.9 to 89.2]
  B Victoria: number analyzed (Participants) | 470 | 483
  B Victoria | 87.2 [83.9 to 90.1] | 88.6 [85.4 to 91.3]
  B Yamagata: number analyzed (Participants) | 474 | 488
  B Yamagata | 87.8 [84.5 to 90.6] | 91.2 [88.3 to 93.5]
Statistical Analysis 1: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For A/H1N1 strain, difference in SCR was defined as SCR after 0.5-mL dose(s) of Fluzone Quadrivalent Vaccine minus SCR after 0.25-mL dose(s) of Fluzone Quadrivalent Vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference in SCRs was >-10%; Difference in SCR (A/H1N1) = 5.1, 95% CI 2-sided [0.189 to 10.0] — A/H1N1 strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)
Statistical Analysis 2: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For A/H3N2 strain, difference in SCR was defined as SCR after 0.5-mL dose(s) of Fluzone Quadrivalent Vaccine minus SCR after 0.25-mL dose(s) of Fluzone Quadrivalent Vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference in SCRs was >-10%; Difference in SCR (A/H3N2) = 4.3, 95% CI 2-sided [-0.283 to 8.99] — A/H3N2 strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)
Statistical Analysis 3: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For B Victoria lineage strain, difference in SCR was defined as SCR after 0.5-mL dose(s) of Fluzone Quadrivalent Vaccine minus SCR after 0.25-mL dose(s) of Fluzone Quadrivalent Vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference in SCRs was >-10%; Difference in SCR (B Victoria lineage) = 1.4, 95% CI 2-sided [-2.78 to 5.56] — B Victoria lineage strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)
Statistical Analysis 4: Comparison: Fluzone Quadrivalent Vaccine, 0.25-mL vs Fluzone Quadrivalent Vaccine, 0.5-mL; For B Yamagata lineage strain, difference in SCR was defined as SCR after 0.5-mL dose(s) of Fluzone Quadrivalent Vaccine minus SCR after 0.25-mL dose(s) of Fluzone Quadrivalent Vaccine; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference in SCRs was >-10%; Difference in SCR (B Yamagata lineage) = 3.4, 95% CI 2-sided [-0.465 to 7.36] — B Yamagata lineage strain: Fluzone Quadrivalent Vaccine (0.5-mL vs. 0.25-mL)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to Day 28 post-final vaccination.
Description: All AEs were presented.
Arm/Group | Fluzone Quadrivalent Vaccine, 0.25-mL | Fluzone Quadrivalent Vaccine, 0.5-mL
All-Cause Mortality (participants affected / at risk) | 0/949 | 0/992
Serious Adverse Events (participants affected / at risk) | 5/949 | 5/992
Other Adverse Events (participants affected / at risk) | 698/949 | 737/992
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone Quadrivalent Vaccine, 0.25-mL (N=949) | Fluzone Quadrivalent Vaccine, 0.5-mL (N=992)
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone Quadrivalent Vaccine, 0.25-mL (N=949) | Fluzone Quadrivalent Vaccine, 0.5-mL (N=992)
Diarrhoea (Gastrointestinal disorders) | 54 | 58
Vomiting (Gastrointestinal disorders) | 115 | 109
Crying (General disorders) | 302 | 321
Injection site erythema (General disorders) | 210 | 228
Injection site pain (General disorders) | 430 | 473
Injection site swelling (General disorders) | 117 | 138
Pyrexia (General disorders) | 151 | 164
Upper respiratory tract infection (Infections and infestations) | 69 | 70
Decreased appetite (Metabolism and nutrition disorders) | 249 | 267
Somnolence (Nervous system disorders) | 292 | 294
Irritability (Psychiatric disorders) | 431 | 458
Cough (Respiratory, thoracic and mediastinal disorders) | 109 | 107
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 74 | 74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT02915302/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT02915302/SAP_001.pdf